CLINICAL TRIAL: NCT00557388
Title: Dietary Strategies to Promote Muscle Protein Anabolism in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: National Nutrition and Food Technology Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MEC 07-3-086; TIFN A-1002
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Sarcopenia
Keywords: muscle loss; aging; protein; amino acids; exercise; protein synthesis
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Motor Activity | interventions — Proteins; Amino Acids; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- 1 (Experimental): Young men 18-30 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids; Other: Physical exercise
- 2 (Experimental): Young men 18-30 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids
- 3 (Experimental): Old men 70-85 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids; Other: Physical exercise
- 4 (Experimental): Old men 70-85 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids
- 5 (Experimental): Old men 70-85 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids
- 6 (Experimental): Old men 70-85 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids
- 7 (Experimental): Old men 70-85 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids
- 8 (Experimental): Old men 70-85 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids
- 9 (Experimental): Old men 70-85 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids
- 10 (Experimental): Old men 70-85 years, BMI < 27 kg/m2
  Interventions: Dietary Supplement: Protein/Amino Acids

INTERVENTIONS:
Dietary Supplement: Protein/Amino Acids — Casein Whey Leucine
Other: Physical exercise — The physical exercise protocol will consist of low intensity cycling and light resistance-type exercise; after 5 minutes of self-paced cycling, subjects will perform 6 sets of 10 repetitions on the horizontal leg press machine (Technogym BV, Rotterdam, The Netherlands) and 6 sets of 10 repetitions on the leg extension machine (Technogym BV, Rotterdam, The Netherlands). The first 2 sets of both resistance exercises will be performed at 40% of the subjects' 1RM. Sets 3-4, and 5-6 will be performed at 55% and 75% of 1RM, respectively, with 2 minutes rest intervals between sets.
  Arms: 1; 3

SUMMARY:
Aging is associated with the loss of lean muscle mass, termed sarcopenia. Food intake and in particular the ingestion of protein or amino acids has been shown to be a powerful stimulus to promote net muscle protein anabolism. However this anabolic response following a meal-like protein bolus seems to be blunted in the elderly as compared to young adults.

The first aim of this proposal is to investigate the post-prandial muscle protein synthesis rates in young and elderly men in response to a meal-like protein bolus after a period of rest or physical activity (study A). The rest trial (REST) will act as a proof-of-principle study to examine the blunted protein synthetic response in the elderly, and as a control trial in comparison with the exercise trial (EXC) to establish the surplus value of physical activity prior to protein intake on muscle protein synthesis.

The second aim of this proposal is to determine the surplus value of an increased quantity of the ingested protein bolus (study B). Large amounts of protein (40 and 60 g) will be compared to a meal-like amount of protein (20 g) as a means to maximize plasma amino acid availability and/or to stimulate muscle protein anabolism.

The third aim of this proposal is to study the differences in quality of the ingested protein bolus (study C). Instead of significantly increasing the quantity of the protein bolus, we will also apply a more practical approach to augment skeletal muscle protein synthesis rates; modifying the digestibility or amino acid composition of a meal-like protein bolus.

ELIGIBILITY:
Inclusion Criteria:

* In study A, non-obese male subjects (BMI <27) between the age of 18-30 yrs and 70-85 yrs will be selected.
* In studies B and C, non-obese male subjects (BMI <27) between the age of 70-85 yrs will be selected.

Exclusion Criteria:

* Type II diabetes or other known diseases
* Use of medication
* Female
* Other ages or BMI than indicated above
* Participation in any regular exercise program.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
All interventions will affect muscle protein synthesis. With the application of amino acid tracer methodology we are able to determine muscle protein synthesis. | 6 hours

SECONDARY OUTCOMES:
Differences in rate of uptake/absorption from the intestine. | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Phd, Principal Investigator — Maastricht University
Locations (1):
- University of Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356
- [Derived] Pennings B, Groen B, de Lange A, Gijsen AP, Zorenc AH, Senden JM, van Loon LJ. Amino acid absorption and subsequent muscle protein accretion following graded intakes of whey protein in elderly men. Am J Physiol Endocrinol Metab. 2012 Apr 15;302(8):E992-9. doi: 10.1152/ajpendo.00517.2011. Epub 2012 Feb 14. PMID 22338070
- [Derived] Pennings B, Boirie Y, Senden JM, Gijsen AP, Kuipers H, van Loon LJ. Whey protein stimulates postprandial muscle protein accretion more effectively than do casein and casein hydrolysate in older men. Am J Clin Nutr. 2011 May;93(5):997-1005. doi: 10.3945/ajcn.110.008102. Epub 2011 Mar 2. PMID 21367943
- [Derived] Pennings B, Koopman R, Beelen M, Senden JM, Saris WH, van Loon LJ. Exercising before protein intake allows for greater use of dietary protein-derived amino acids for de novo muscle protein synthesis in both young and elderly men. Am J Clin Nutr. 2011 Feb;93(2):322-31. doi: 10.3945/ajcn.2010.29649. Epub 2010 Nov 17. PMID 21084649